CLINICAL TRIAL: NCT00679510
Title: Phase 2: Effects of Rosuvastatin on Surrogate Markers for Cardiovascular Events in Patients With Rheumatoid Arthritis
Brief Title: Rosuvastatin in Rheumatoid Arthritis (RORA)
Acronym: RORA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21726/0204/001-0001; 2004-001909-10
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Rosuvastatin; Cardiovascular; Intima media thickness
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients were randomly allocated either rosuvastatin (crestor) 10 mgs or placebo. The drugs (rosuvastatin and placebo) were provided by Astra Zeneca Ltd. Computerised randomisation was done by an independent person from Tayside pharmacy and both patients and doctors were unaware of drug allocation. In order to blind the trial drugs during the study period, the blood tests for cholesterol were checked by research nurse who was not involved in the clinical assessment of patients.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rosuvastatin (Active Comparator): Rosuvastatin Patients were randomly allocated rosuvastatin (crestor) 10 mgs. The drugs (rosuvastatin and placebo) were provided by Astra Zeneca Ltd.
  Interventions: Drug: rosuvastatin
- Placebo (Placebo Comparator): Placebo. Patients were randomly allocated placebo. The drugs (rosuvastatin and placebo) were provided by Astra Zeneca Ltd.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rosuvastatin — tablet 10 mgs once daily
  Other Names: crestor
  Arms: rosuvastatin
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
Patients with rheumatoid arthritis are at increased risk of having cardiovascular deaths. The investigator's study is aimed at looking at the effects of proven cholesterol lowering treatment drug called rosuvastatin in rheumatoid arthritis patients on few cardiovascular markers. Endothelial behaviour improved on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be selected from a high risk population of hospital clinic attendees, defined as RA greater than 5 years' disease duration, and all will be RA latex seropositive or IgM RF ELISA >14iu/ml. The subjects will be of either sex and >40 years of age.
* Patients should have both tender and swollen joint counts >4 each and either a CRP >10mg/l, ESR >25mm/h or PV >1.78.
* Patients on cyclosporine or other medications known to be contraindicated with this form of drug will not be enrolled.

Exclusion Criteria:

* The patient's hospital and general practice records will be scrutinised for evidence of symptomatic vascular disease.
* Any patient not free from vascular disease symptoms will be excluded.
* In addition to evidence of symptomatic vascular disease (either previous or current), the exclusion criteria consist also of those already taking lipid-lowering therapy or those with contraindications to these therapies.
* Also excluded will be subjects with a total cholesterol level of >7.5mmol/L as it might be argued that such patients merit primary prevention on the basis of dyslipidemia alone.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
measurement of intima media thickness | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jill Belch, MD FRCP, Study Chair — University of Dundee
Locations (1):
- University of Dundee, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar P, Kennedy G, Khan F, Pullar T, Belch JJ. Rosuvastatin might have an effect on C-reactive protein but not on rheumatoid disease activity: Tayside randomized controlled study. Scott Med J. 2012 May;57(2):80-3. doi: 10.1258/smj.2012.012004. PMID 22555227